CLINICAL TRIAL: NCT06675617
Title: A Clinical Study to Evaluate the Effectiveness and Safety of the Allay® Aortic Stent as Adjunctive Endovascular Treatment of Type B Aortic Dissection in Patients Eligible for Thoracic Endovascular Repair With Stent Grafts
Brief Title: EXtensive mulTilayer stEnt treatmeNt in Aortic disSectiOn
Acronym: EXTENSO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Intressa Vascular SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-P3-03-001
Record Dates: First submitted 2024-10-30; First posted 2024-11-05 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Type B Aortic Dissection
Keywords: TBAD; Allay; aortic; dissection; type B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allay Aortic Stent (Experimental): A covered thoracic stent graft is first deployed in supraceliac position as per standard of care then followed by the implantation of the Allay® Aortic Stent deployed from within the stent graft, extending below the celiac trunk to the end of the dissected aorta, typically the aortoiliac bifurcation.
  Interventions: Device: Allay Aortic Stent

INTERVENTIONS:
Device: Allay Aortic Stent — Endovascular treatment of an aortic dissection

SUMMARY:
This clinical trial is a prospective, multicenter, open label study designed to evaluate the effectiveness and the safety of the Allay® Aortic Stent as adjunctive endovascular treatment of Type B aortic dissection in patients eligible for thoracic endovascular aortic repair with stent grafts.

DETAILED DESCRIPTION:
Thoracic endovascular repair (TEVAR) with stent grafts is recommended for patients with acute complicated or high-risk type B aortic dissection (TBAD) as part of standard of care per current medical guidelines. Although the benefits of TEVAR with stent grafts are well established, there remains a significant risk of late complications, including aortic growth requiring reinterventions, or progression and/or rupture.

In the present clinical investigation, the investigational procedure of adjunctive thoracic stent graft extension with the Allay® Aortic Stent will consist of the placement of a CE-marked Thoracic Stent Graft in the descending thoracic aorta (proximal to the celiac trunk) followed by the implantation of the Allay® Aortic Stent as adjunctive treatment of TBAD.

The study objective is to demonstrate that the Allay® Aortic Stent, used as adjunctive endovascular treatment of Type B aortic dissection in patients eligible for thoracic endovascular aortic repair with stent grafts, results in a low rate of aortic growth requiring secondary reintervention, including open conversion, or aortic rupture in the treated abdominal segment at 12 months. The study will also allow to evaluate the incidence of Major Adverse Events (MAE) following TEVAR, at 30 days post-implantation of the Allay® Aortic Stent.

Based on available data on similar devices, the objective performance goal is set to an expected proportion of 85% freedom from aortic growth requiring secondary reintervention or aortic rupture of the abdominal segment at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Have a type B aortic dissection extending to the celiac trunk or beyond
* Are eligible for thoracic endovascular treatment with stent grafts as per local guidelines, and physician's decision
* Have been elected for treatment with commercially available stent graft as per their IFU within 90 days of dissection symptoms onset

Exclusion Criteria:

* General Exclusion Criteria:

  * Age < 18 years
  * Pregnant, breast-feeding or planning on becoming pregnant during the entire duration of the study
  * Unable to provide written informed consent
  * Unable or unwilling to comply with the requirements of the study protocol
  * Taking part already in an investigational device or drug study that could interfere with the outcomes being studied
  * Active drug addiction or known history of drug abuse within one year of treatment
* Medical Exclusion Criteria:

  * Aortic rupture, free or contained including haemothorax, increasing periaortic hematoma, or mediastinal hematoma
  * Aortic fistula
  * Suspicion of bowel necrosis or irreversible visceral ischemia
  * Stage 5 chronic kidney disease
  * Life expectancy of less than 2 years due to any other medical condition than the dissection to be treated
  * Active malignancy
  * Known sensitivities or allergies to the device materials (including cobalt, chromium, nickel)
  * Known sensitivities or allergies to contrast materials that cannot be pre-medicated
  * Mycotic aortic aneurysm or active systemic infection that may place the patient at increased risk of endovascular infection
  * American Society of Anaesthesiologists (ASA) class V (moribund patient not expected to live 24 hours with or without operation)
  * Diagnosed or suspected congenital degenerative connective tissue disease (e.g., Marfan's, Loeys-Dietz or Ehlers-Danlos syndrome)
  * Uncorrectable coagulopathy, bleeding diathesis or refusal of blood transfusion
  * Any major cardiovascular or cerebrovascular ischemic event, including myocardial infarction or stroke, or treatment of such event, within 90 days prior to enrolment
  * Any aortic-related interventional or surgical procedure within 30 days prior to enrolment
  * Any planned aortic-related interventional or surgical procedure within 30 days after the study procedure
* Anatomical Exclusion Criteria:

  * Aneurysmal dilatation of the false lumen defined as maximum transaortic diameter >55 mm in women or >60 mm in men in the thoraco-abdominal segment or >50 mm in women or >55 mm in men in the abdominal segment, measured inner-wall to inner-wall;
  * Inadequate proximal landing zone for the stent graft, such zone being <20 mm long
  * Inadequate proximal landing zone geometry for the Allay® Aortic Stent (e.g. aortic kink)
  * Planned implantation of a stent graft with a distal diameter >38 mm or <20 mm
  * Aorta or iliac anatomy not allowing the advancement of the delivery system
  * Subject in whom the thoracic stent graft is either 1) not implanted in its intended position and/or 2) leads to any serious device complication, and/or who has 3) persistent static obstruction of the visceral or both renal arteries, prior to Allay® Aortic Stent implantation, will not be implanted with the Allay® Aortic Stent and will be withdrawn from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Freedom from aortic growth requiring secondary reintervention, including open conversion, or aortic rupture in the region treated by the Allay® Aortic Stent at 12 months | 12 months
  An aortic growth requiring reintervention in the region treated with the Allay® Aortic Stent is defined as an increase in maximum aortic transverse diameter >10mm at 12 months relative to the first post-operative CT scan done at discharge and not later than 30 days.

SECONDARY OUTCOMES:
Percentage of Participants with Successful Technical Performance of the Allay® Aortic Stent Implantation | At index procedure
  Technical success of the implantation of the Allay® Aortic Stent will be assessed at index procedure as the composite endpoint of the following:
  * Successful delivery to the intended implantation site and withdrawal of the delivery system;
  * Accurate deployment of the Allay® Aortic Stent defined as appropriate proximal landing in the stent graft and distal landing in descending aorta;
  * Absence of unexpected adverse effect on the stent graft, additional procedure related to the device, procedure, or withdrawal of the delivery system.
Incidence of Major Adverse Events (MAE) within 30 Days After Allay® Aortic Stent Implantation | 30 days
  The safety endpoint will be assessed as the freedom from Major Adverse Events (MAE) at 30 days, defined as the composite endpoint of the following new-onset adverse events:
  * Myocardial infarction;
  * Renal failure requiring permanent dialysis;
  * Bowel ischemia requiring surgical intervention;
  * Disabling stroke;
  * Paraplegia or paraparesis;
  * Limb ischemia;
  * Death.
Freedom from all-cause mortality; | Immediately at discharge and subsequent follow-up visits, at 30 days, 12, 24, 36, 48 and 60 months
  The percentage of patients alive from any cause post-discharge at follow-up intervals.
Freedom from Dissection-Related Mortality | Immediately at discharge and subsequent follow-up visits at 30 days, 12, 24, 36, 48, and 60 months.
  The percentage of patients who are alive and free from dissection-related mortality, if known.
Freedom from Readmission (Post-Discharge) | Subsequent follow-up visits at 30 days, 12, 24, 36, 48, and 60 months.
  The percentage of patients who have not been readmitted to the hospital post-discharge.
Freedom from Aorta-Related Reintervention | Immediately at discharge and subsequent follow-up visits at 30 days, 12, 24, 36, 48, and 60 months.
  The percentage of patients who have not required a reintervention related to the aorta, including details on the type and frequency if any.
Freedom from Open Conversion | Immediately at discharge and subsequent follow-up visits at 30 days, 12, 24, 36, 48, and 60 months.
  The percentage of patients who have not required conversion to open surgical intervention.
Freedom from New Ischemia | Immediately at discharge and subsequent follow-up visits at 30 days, 12, 24, 36, 48, and 60 months.
  The percentage of patients free from new ischemic events identified post-intervention.
Freedom from Reintervention Related to Side Branches | Immediately at discharge and subsequent follow-up visits at 30 days, 12, 24, 36, 48, and 60 months.
  The percentage of patients who have not required reintervention related to side branches.
Aortic rupture | Assessed at discharge or not later than 30 days from index procedure, and then compared to pre-operative CT scan
  Incidence of aortic rupture observed through CT imaging post-intervention.
Percentage of Participants with Patent Major Aortic Branches Post-Allay® Aortic Stent Implantation | Assessed at discharge (or within 30 days from the index procedure) and compared to the pre-operative CT scan.
  Assessment of changes in the patency of major aortic branches post-intervention.
Percentage of Participants with Patent Major Descending Aortic Branches Covered by the Allay® Aortic Stent | Assessed at discharge (or within 30 days from the index procedure) and compared to the pre-operative CT scan.
  Evaluation of changes in the patency of major descending aortic branches covered by the Allay® Aortic Stent.
Percentage of Participants with Device Deficiencies Detected by CT Imaging Post-Allay® Aortic Stent Implantation | Assessed at discharge (or within 30 days from the index procedure) and compared to the pre-operative CT scan.
  Assessment of device deficiencies observed through CT imaging, including loss of patency, kink, collapse, migration, and overlap separation.
Aortic growth | Assessed at 12, 24, 36, 48 and 60 months, then compared to first post-operative CT scan done at discharge and not later than 30 days from index procedure
  Measurement of aortic growth over time as assessed through CT imaging.
Aortic Rupture | Assessed at 12, 24, 36, 48, and 60 months, compared to the first post-operative CT scan done at discharge.
  Incidence of aortic rupture observed during follow-up CT imaging.
New Dissection or Extension of Dissection | Assessed at 12, 24, 36, 48, and 60 months, compared to the first post-operative CT scan.
  Occurrence of any new dissection or extension of existing dissection observed in follow-up CT scans.
Percentage of Participants with Fistula Formation Detected on Follow-Up CT Imaging | Assessed at 12, 24, 36, 48, and 60 months, compared to the first post-operative CT scan.
  Identification of fistula formation during follow-up CT imaging assessments.
Change in True Lumen, False Lumen, and Transaortic Diameters | Assessed at 12, 24, 36, 48, and 60 months, compared to the first post-operative CT scan.
  Measurement of changes in the true lumen, false lumen, and transaortic diameters through follow-up CT imaging.
Percentage of Participants with Maintained Patency in Major Aortic Branches on Follow-Up Imaging | Assessed at 12, 24, 36, 48, and 60 months, compared to the first post-operative CT scan.
  Evaluation of changes in the patency of major aortic branches during follow-up imaging.
Percentage of Participants with Maintained Patency in Major Descending Aortic Branches Covered by the Allay® Aortic Stent on Follow-Up Imaging | Assessed at 12, 24, 36, 48, and 60 months, compared to the first post-operative CT scan.
  Observation of changes in the patency of major descending aortic branches covered by the Allay® Aortic Stent.
Percentage of Participants with Maintained False Lumen Perfusion and Patency in All Treated Segments on Follow-Up Imaging | Assessed at 12, 24, 36, 48, and 60 months, compared to the first post-operative CT scan.
  Assessment of false lumen perfusion and patency across all treated segments.
Percentage of Participants with Device Deficiencies on Follow-Up Imaging | Assessed at 12, 24, 36, 48, and 60 months, compared to the first post-operative CT scan.
  Identification of device deficiencies through CT imaging, including but not limited to stent integrity, patency loss (kink, collapse), migration, separation, and endoleak Types I or III.

CONTACTS AND LOCATIONS:
Overall Officials: Wolf-Hans Eilenberg, MD, PhD, FEBVS, Principal Investigator — Medical University of Vienna
Locations (10):
- Belgium (3):
  - Ziekenhuis Oost-Limburg, Genk
  - UZ Leuven, Leuven
  - CHU Liège, Liège
- Acibadem City Clinic University Hospital and Cardiovascular Center, Sofia, Bulgaria
- Hopital Européen Georges Pompidou AP-HP, Paris, France
- Germany (3):
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Universitätsklinikum Leipzig AöR, Leipzig
  - University Hospital of Münster, Münster
- University Clinical Centre of Serbia, Belgrade, Serbia
- Republican Research Centre of Emergency Medicine, Tashkent, Uzbekistan

IPD SHARING:
Plan to Share IPD: Undecided